CLINICAL TRIAL: NCT06961565
Title: A Phase 1/1b Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of PAS-004, a MAPK/ERK Kinase 1/2 (MEK 1/2) Inhibitor, in Adult Participants With Neurofibromatosis Type 1 (NF1) With Symptomatic and Inoperable, Incompletely Resected, or Recurrent Plexiform Neurofibromas
Brief Title: PAS-004 in Adults Who Have Neurofibromatosis Type 1 With Plexiform Neurofibromas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pasithea Therapeutics Corp. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PAS-004-103
Record Dates: First submitted 2025-04-11; First posted 2025-05-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: NF1 Mutation; Neurofibroma Plexiform; Neurofibroma, Plexiform; Neurofibromatosis Type 1 (NF1)-Related Plexiform Neurofibromas (PNs); Neurofibromatosis Type 1 (NF1)
Keywords: NF1; neurofibromatosis; plexiform neurofibroma; cutaneous neurofibroma; neurofibromatosis type 1
MeSH Terms: conditions — Neurofibroma, Plexiform; Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Intervention Model Description: 3+3 dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Sequential dose escalation: 4 mg, 8 mg, 12 mg, and 18 mg
  Interventions: Drug: PAS-004 Tablets
- Part B (Experimental): Two parallel cohorts dosing at 2 levels selected based on Part A safety results
  Interventions: Drug: PAS-004 Tablets

INTERVENTIONS:
Drug: PAS-004 Tablets — A mitogen-activated protein kinase/extracellular signal-regulated kinase kinase (MAPK/ERK kinase, or MEK) 1/2 inhibitor presented in 1m and 4mg strength tablets, intended for oral administration once daily.

SUMMARY:
The main purpose of this clinical trial is to test PAS-004 in people with at least one symptomatic plexiform neurofibroma due to Neurofibromatosis Type 1 (NF1). The main questions it aims to answer are:

* How well participants are able tolerate different doses of PAS-004, and
* What side effects PAS-004 might have.

This study will have two parts, Part A and Part B. The main goal of Part A of this study is to learn more about how participants tolerate different doses of PAS-004, and what side effects PAS-004 might have. What we learn from Part A of the study will help decide what doses of the study drug (PAS-004) should be used in Part B of the study, and if it is safe.

In Part B, two different doses from Part A will be tested. The main goal of this part of the study is to keep studying any side effects of PAS-004 at those two dose levels, and to learn more about if the doses picked for this part of the study might have an effect on plexiform neurofibromas.

Participants in Part A of the study who were taking doses selected for Part B may be able to continue on to Part B and keep taking the same dose of PAS-004 for 6 more months.

Study participants in both parts will have regular visits to the study doctor and be asked to have tests and exams done to check on their health and safety, including blood draws and MRIs. Everyone participating in the study will take PAS-004 by mouth once a day during the study, in 28-day cycles. Participants will be asked to keep a diary to record their daily dose of study drug.

Participants will continue on daily PAS-004 for up to 6 months, or until:

* They decide to withdraw from the study, or
* They experience unacceptable side effects, or
* Their disease progresses, or another illness interferes with taking the study drug, or
* The sponsor selects a dose level to study further in the next part of the study, or
* The sponsor stops the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is capable of providing informed consent, which includes compliance with the requirements, prohibitions and restrictions listed in the informed consent form.
2. Participant has been informed both verbally and in writing about the objectives of the clinical study, the methods, the anticipated benefits, the potential risks, and the discomfort to which they may be exposed and has given written consent to participation in the study prior to study start and any study-related procedure.
3. Participant must be at least 18 years of age at the signing of the informed consent form (ICF).
4. Participant must be able to swallow oral medication.
5. Performance status: Participant must have a Karnofsky performance level of ≥70%. Note: Participants who are wheelchair bound because of paralysis secondary to a PN should be considered ambulatory when they are in the wheelchair. Similarly, participants with limited mobility secondary to the need for mechanical support (such as an airway PN requiring tracheostomy or CPAP) will also be considered ambulatory for the purposes of this study.
6. Participant has been diagnosed with NF1 based upon the following diagnostic criteria:

   a. Clinical and imaging confirmation meeting at least two of the following NF1 diagnostic criteria in accordance with the clinical NIH consensus criteria: i. ≥ Six cafe-au-lait macules > 1.5 cm in maximum diameter ii. Axillary and/or inguinal freckling iii. ≥ Two neurofibromas of any type, or ≥ 1 plexiform neurofibroma; iv. An optic pathway glioma (prior diagnosis without concurrent disease is acceptable) v. ≥ Five Lisch nodules (iris hamartomas). Note: must be confirmed on slit lamp exam by an ophthalmologist if this is one of only two criteria met for diagnosis vi. A distinctive bony lesion such as dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex vii. Biologic parent with confirmed diagnosis of NF1 viii. Genetic testing demonstrating a pathogenic NF1 germline mutation per CLIA-certified laboratory (or equivalent) testing.

1. Note: NF1 germline pathologic mutation positive must either be confirmed by the central laboratory or have documentation of NF1 mutation issued by a CLIA-certified laboratory (or equivalent). 2. No concern by the Investigator that an NF1 mimic, including but not limited to Noonan Syndrome, Legius Syndrome, or schwannomatosis could potentially serve as a more likely diagnosis

7. Participants satisfying the NF1 diagnostic criteria outlined in Inclusion Criterion #6 must also meet one of the following criteria:

a. Participant has at least one symptomatic PN ("Target PN") measuring at least 3 cm on maximal cross-sectional (axial) diameter that is judged by the Investigator to be likely responsible for participant symptoms (such as pain, deformity, or neurologic disability), and unable to be completely resected without causing substantial damage/functional deficit, or unsuitable for surgery with high surgical risks.

b. Participant has an incompletely resected symptomatic PN with a postoperative residual of at least 15% of the primary lesion and measuring at least 3 cm on cross-sectional (axial) diameter.

c. Participant has a recurrent symptomatic PN measuring at least 3 cm in maximal cross-sectional (axial) dimension after prior resection.

8. Participants should have a minimum of seven measurable CN measuring 6-15 mm (if participants satisfy Inclusion Criterion #6 and have no CN or less than 7 CN they still might be considered for the study as judged by the Investigator and Sponsor).

1. Measurable is defined as: 1. non-pedunculated (no stalk) 2. surrounded by visually uninvolved skin and not in physical contact with another CN, 3. measuring between 6 and 15 mm in the longest diameter and exophytic on visual exam (not macular).
2. At least seven CN should be located on the trunk, neck, and/or limbs measuring between 6 and 15 mm in maximal diameter, and "measurable" as per the definition listed above.
3. Participants with CN meeting the above criteria will undergo optional resections of at least two CN that meet eligibility criteria. If participant is willing to accept additional CN resections, this is permitted for up to four additional lesions after completion of six PAS-004 treatment cycles or after early withdrawal as long as there are sufficient lesions to allow efficacy assessment.

   9. Participant must be able and willing to undergo serial MRI scans as outlined in the study protocol.

   Note: Anxiolytic medication or pain medication as deemed clinically appropriate by the Investigator is permissible for the purposes of managing anxiety, claustrophobia, and pain during MRI.

   10. Participant must be able and willing to undergo serial 2-D and where available 3-D photography as well as caliper measurements as outlined in the study protocol.

   11. Participant must have an international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 x ULN.

   12. Participant must have adequate organ and bone marrow function at screening as indicated by the following laboratory value ranges:

a. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L b. Hemoglobin ≥ 90 g/dL c. Platelets ≥ 100 × 109/L d. Serum total bilirubin ≤ 1.5 × ULN for age (≤ 3.0 × ULN in participants with Gilbert's syndrome) e. Serum total bilirubin ≤ 1.5 × ULN (Serum total bilirubin can be ≤ 3.0 × ULN if participants have hemolysis or congenital hemolytic diseases) f. Aspartate aminotransferase (AST) ≤ 2.0 × ULN g. Alanine aminotransferase (ALT) ≤ 2.0 × ULN h. Albumin ≥ 3 g/dL i. Creatinine clearance ≥ 60 mL/min

13. Participant must either agree to maintain abstinence (no heterosexual intercourse), or to use one highly effective form of contraception during study treatment and for at least 90 days after the last dose of investigational product (IP). Sperm-producing participants must agree not to donate sperm while receiving IP and for at least 90 days after the last dose of IP.

Exclusion Criteria:

1. Participant has participated in another interventional clinical study within 28 days of starting PAS-004.
2. Participant has received chemotherapy for any indication within 90 days of starting PAS-004.
3. Participant has ongoing side effects from prior chemotherapy that are worse than mild (except alopecia). ("Mild" is defined as Asymptomatic or mild symptoms, clinical or diagnostic observations only, or intervention not indicated.)
4. Participant has received treatment with any PN-directed drug or biologic therapy within 14 days of starting PAS-004.
5. Participant has received treatment with a strong CYP3A4 inhibitor or inducer, or moderate inducers for CYP2C8 and CYP2C9 within 14 days of starting PAS-004, or any drug considered a major substrate of the enzymes above with a narrow therapeutic index except for topical skin use, as judged by the Investigator and Sponsor.
6. Participant has received growth factors to increase the number or function of platelets or white blood cells within 7 days of starting PAS-004.
7. Participant has received radiotherapy, major surgery, or immunotherapy within 28 days of starting PAS-004.
8. Participant has malignant tumors associated with NF1 requiring chemotherapy, radiotherapy, or surgery, such as intermediate- to high-grade gliomas or malignant peripheral nerve sheath tumors.
9. Participant has a current malignancy (excluding cured non-melanomatous skin cancer, breast carcinoma in situ, or cervical cancer in situ) or has history of malignancy requiring active treatment within the past 5 years (excluding cured non-melanomatous skin cancer, breast carcinoma in situ, and cervical cancer in situ). Other tissue-limited low stage cancers can be assessed by the Sponsor for possible inclusion on a per-participant basis.
10. Participant has uncontrolled hypertension defined as blood pressures >150/90 mmHg on repeat examinations despite maximal medical management.

    Note: Participants with controlled hypertension with anti-hypertension therapy are permitted, as judged by the Investigator and Sponsor.
11. Participant has active dysphagia, digestive system disease, malabsorption syndrome, or other conditions that might affect the absorption of PAS-004.
12. Participant has previous or current retinal vein occlusion (RVO), retinal pigment epithelial detachments (RPED), clinically active glaucoma, or other significant abnormality in screening ophthalmic examination.
13. Participant has interstitial pneumonia, NF1-related pulmonary disease, including existing clinically significant radiation pneumonitis.
14. Participant has impaired cardiac function or cardiac disease as indicated by:

    1. Average QTc interval > 480 ms calculated using the Fridericia's QT interval correction formula.
    2. Grade ≥ 3 congestive heart failure per New York Heart Association (NYHA) guidelines.
    3. Clinically significant arrhythmias, including but not limited to, complete left bundle branch conduction abnormalities and 2nd degree atrioventricular block.
    4. Known concurrent clinically significant coronary artery disease, cardiomyopathy, or severe valvular disease.
    5. Echocardiogram or multi-gated acquisition (MUGA) scan performed during the screening showing impaired left ventricular ejection fraction (LVEF) < 45%.
15. Participant has taken a QTc-prolonging medication within seven days of IP initiation or longer if the half-life of the QTc prolonging medication is such that the drug is not cleared from the body within 7 days (5 half-lives) of IP initiation.
16. Participant has an uncontrolled bacterial, fungal, or viral infections, including active hepatitis B (hepatitis B virus surface antigen positive and hepatitis B virus DNA > 1000 IU/ml or meeting the study site's diagnostic criteria for active hepatitis B infection), hepatitis C (hepatitis C virus RNA positive), or human immunodeficiency virus (HIV) infection with detectable viral load.
17. Any clinically significant active or known history of liver disease or known hepatobiliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
18. Participant has a known hypersensitivity to PAS-004, its excipients, or another MEK 1/2 inhibitor.
19. Participant is pregnant or lactating.
20. Participant has a clinically significant condition that, in the opinion of the investigator, would preclude study participation or compliance with safety requirements.
21. Participant is unable to attend in-person clinic visits per clinical site guidelines and restrictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Part A: To evaluate the safety and tolerability of PAS-004 when administered for one 28-day treatment cycle | Part A from enrollment (Day 1) through Day 28 (completion of Cycle 1)
  Endpoint/Outcome Measures:
  Number of participants with dose-limiting toxicities (DLTs), with Adverse Events (AEs), AEs leading to interruption or discontinuation of study drug, with clinically significant findings on clinical laboratory tests, with abnormal cardiac and visual function exams using the Common Terminology Criteria for Adverse Events (CTCAE Version 5).
Part B: To evaluate the safety and tolerability of PAS-004 when administered for six 28-day treatment cycle | Part B from enrollment (Day 1) through Day 168 (completion of Cycle 6) [each cycle is 28 days]
  Endpoint/Outcome Measures:
  Number of participants with dose-limiting toxicities (DLTs), with Adverse Events (AEs), AEs leading to interruption or discontinuation of study drug, with clinically significant findings on clinical laboratory tests, with abnormal cardiac and visual function exams using the Common Terminology Criteria for Adverse Events (CTCAE Version 5).

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day 28 (predose, and 1 , 3 , 6 , and 24 hours post-dose) [end of Cycle 1]
Plasma predose or trough concentration (Ctau/Ctrough) | Day 28 (predose, and 1 , 3 , 6 , and 24 hours post-dose) [end of Cycle 1]
Time of maximum plasma concentration (Tmax) | Day 28 (predose, and 1 , 3 , 6 , and 24 hours post-dose) [end of Cycle 1]
Area under the concentration versus time curve for the dosing interval, assuming steady state has been reached and duplicating the predose concentration for the 24 hour postdose concentration (AUC0-tau) | Day 28 (predose, and 1 , 3 , 6 , and 24 hours post-dose) [end of Cycle 1]
Evaluation of the percentage of extracellular signal-regulated kinase phosphorylation (pERK) inhibition from baseline | Day 1 through Day 28 (Cycle 1), and at each subsequent 28-day cycle through Cycle 6 (D168) [each cycle is 28 days]
  Analysis of pERK inhibition will be performed on peripheral blood mononuclear cells (PBMCs).
Evaluation of the clinical benefit rate (CBR) over time on MRI with volumetric analysis of plexiform neurofibroma(s) using Response Evaluation in Neurofibromatosis and Schwannomatosis (REiNS) criteria | Screening (Baseline), Day 112 (End of Cycle 4), and Day 168 (End of Cycle 6) [each cycle is 28 days]
Evaluation of the best objective response rate (ORR) over time on MRI with volumetric analysis of plexiform neurofibroma(s) using REiNS criteria | Screening (Baseline), Day 112 (End of Cycle 4), and Day 168 (End of Cycle 6) [each cycle is 28 days]
Evaluation of time to maximal response on MRI with volumetric analysis of plexiform neurofibroma(s) using the REiNS criteria | Screening (Baseline), Day 112 (End of Cycle 4), and Day 168 (End of Cycle 6) [each cycle is 28 days]
Evaluation of the appearance of cutaneous neurofibromas over time using photography | Screening (Baseline), Day 112 (End of Cycle 4), and Day 168 (End of Cycle 6) [each cycle is 28 days]
Evaluation of the size of cutaneous neurofibromas over time | Screening (Baseline), Day 112 (End of Cycle 4), and Day 168 (End of Cycle 6) [each cycle is 28 days]
  Cutaneous neurofibromas will be measured by investigators using digital calipers, and centrally on 2D photographs
Evaluation of changes from baseline on quality of life (QOL) using the Plexi-QOL survey | Screening, and Days 28, 56, 84, 112, 140 and 168
  Plexiform neurofibromas Quality of Life measure (PlexiQoL). The PlexiQoL consists of 18 items with a dichotomous response option (True / Not True). The number of times that a participant chooses 'True' is summed to produce a score ranging from 0 to 18, with a higher score indicating poorer QoL.
Evaluation of changes from baseline on any physical symptoms attributed to the target plexiform neurofibroma using the Patient-Reported Outcomes Measurement Information System (PROMIS©) Physical Function (PF) assessment | Screening, and Days 28, 56, 84, 112, 140 and 168
  Patient Reported Outcome Measurement Information System (PROMIS©) Physical Function (PF) assessment (Short Form v2.0 Physical Function 10b). The short form contains 10 questions, and each item is scored on a 5-point rating scale (1 [unable to do] to 5 [without any difficulty]), with higher scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago R Marques, MD, Study Director — Pasithea Therapeutics Corp.
Locations (5):
- University of Alabama at Birmingham, Birmingham, Alabama, United States
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- South Korea (2):
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Sinchŏn-dong

IPD SHARING:
Plan to Share IPD: No